CLINICAL TRIAL: NCT01683435
Title: The Value of Hyaluronic Binding Assays (HBA) in the Evaluation of Idiopathic Infertility
Brief Title: The Value of HBA in the Evaluation of Idiopathic Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 11-134
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hylauronin binding assay (Experimental): HBA binding assay will be preformed on the discarded portion of semen analysis used for IVF.
  Interventions: Other: HBA binding assay

INTERVENTIONS:
Other: HBA binding assay — HBA binding assay will be preformed on the discarded portion of semen analysis used for IVF.

SUMMARY:
We would like to determine if HBA® testing of sperm in couples with presumed idiopathic infertility will reveal lower binding percentages than in couples with an identifiable cause of infertility either male factor or tubal factor

DETAILED DESCRIPTION:
We would like to determine if HBA® testing of sperm in couples with presumed idiopathic infertility will reveal lower binding percentages than in couples with an identifiable cause of infertility either male factor or tubal factor We would like to determine if patients with abnormal HBA binding have decreased IVF outcome: decreases clinical pregnancy rate, implantation rate, and increased miscarriage rate

ELIGIBILITY:
Inclusion Criteria:

* . All groups will include females under 40 years of age undergoing 1st IVF cycle 3 groups

  1. Abnormal Semen Analysis (sperm count <10 million/ml and /or rapid progressive motility < 50 %, WHO morphology <30%) normal HSG , normal ovarian reserve testing and ovulation testing
  2. Unexplained infertility- normal ovarian reserve testing and ovulation testing (FSH< 10, AMH>1.0) Normal ovulatory cycles, normal WHO semen analysis. Normal tubes on HSG or Laparoscopy
  3. Tubal infertility as assessed by HSG or laparoscopy

Exclusion Criteria:

* women over 40, prior failed IVF

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
In each of these groups we will assess presence of HBA bound sperm | immediate at time of preforming HBA test

CONTACTS AND LOCATIONS:
Overall Officials: Martin Keltz, MD, Principal Investigator — Mount Sinai St. Luke's
Locations (1):
- The Continuum Reproductive Center, New York, New York, United States